CLINICAL TRIAL: NCT00004754
Title: Phase IV Study of Chronic Infusional Epoprostenol for Severe Primary Pulmonary Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Baylor College of Medicine (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 199/11678; BCM-P1850
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Hypertension, Pulmonary
Keywords: cardiovascular and respiratory diseases; hypertensive disorder; primary pulmonary hypertension; rare disease
MeSH Terms: conditions — Hypertension, Pulmonary; Respiratory Tract Diseases; Hypertension; Familial Primary Pulmonary Hypertension; Rare Diseases | interventions — Epoprostenol

INTERVENTIONS:
Drug: epoprostenol

SUMMARY:
OBJECTIVES: I. Provide epoprostenol (Flolan, prostaglandin I2) by chronic infusion to patients with severe primary pulmonary hypertension for whom no alternative therapy is available.

II. Obtain additional safety information on continuous infusion epoprostenol. III. Obtain additional information on economic resource health consumption.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are treated with a chronic continuous infusion of epoprostenol.

The highest tolerated infusion rate is determined for each patient by gradually increasing the rate until the target dose is reached or the patient experiences at least 1 dose-limiting effect.

Patients are subsequently treated with a chronic continuous infusion, beginning at a rate below the highest tolerated rate. Attempts are made to increase the dose to the highest tolerated rate over the first 72 hours.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

* Severe primary pulmonary hypertension
* Able to prepare and self-administer medication

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-08

CONTACTS AND LOCATIONS:
Overall Officials: Adaani E. Frost, Study Chair — Baylor College of Medicine